CLINICAL TRIAL: NCT01226719
Title: A Phase II Study of FOLFOXIRI Plus Panitumumab Followed by Evaluation for Resection, in Patients With Metastatic KRAS Wild-Type Colorectal Cancer With Liver Metastases Only
Brief Title: FOLFOXIRI Plus Panitumumab Patients With Metastatic KRAS Wild-Type Colorectal Cancer With Liver Metastases Only
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 134
Record Dates: First submitted 2010-10-15; First posted 2010-10-22 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Cancer
Keywords: liver-only metastatic KRAS wild-type colorectal cancer; Panitumumab; Oxaliplatin; Irinotecan; Leucovorin; 5-Fluorouracil
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Combined Modality Therapy; Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFOXIRI+panitumumab regimen (Experimental): All patients will receive the FOLFOXIRI/panitumumab regimen, with drugs administered in the following order:
  * Panitumumab
  * Oxaliplatin
  * Irinotecan
  * Leucovorin
  * 5-Fluorouracil
  Interventions: Drug: Panitumumab; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Panitumumab — 6 mg/kg, 60-90 minute IV infusion every 2 weeks
  Other Names: Combined Modality Treatment
Drug: Oxaliplatin — 85 mg/m2, 2-hour IV infusion every 2 weeks
  Other Names: Combined Modality Treatment
Drug: Irinotecan — 125 mg/m2, 1-hour IV infusion every 2 weeks
  Other Names: Combined Modality Treatment
Drug: Leucovorin — 200 mg/m2, 2-hour IV infusion every 2 weeks
  Other Names: Combined Modality Treatment
Drug: 5-Fluorouracil — 3200 mg/m2 IV, 48-hour continuous infusion every two weeks
  Other Names: Combined Modality Treatment

SUMMARY:
In this Phase II study the investigators plan to determine the overall response rate (ORR) of the combination of FOLFOXIRI plus panitumumab as first-line treatment of patients with liver-only metastatic KRAS wild-type colorectal cancer.

DETAILED DESCRIPTION:
Further data has emerged showing a consistent lack of efficacy using EGFR inhibitor panitumumab in combination with chemotherapy in the treatment of patients with KRAS mutant colorectal cancer. For patients with liver-only metastatic colorectal cancer, improvement in response rates with newer chemotherapy regimens has led to a larger percentage of patients eligible for surgical resection. Treatment with FOLFOXIRI improves response rates when compared to FOLFIRI. Similarly, the addition of an EGFR inhibitor improves the response rate of FOLFIRI in patients with wild-type KRAS. In this trial, we will attempt to maximize the response rate and the surgical resection rate by using FOLFOXIRI and panitumumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a biopsy confirmed adenocarcinoma of the colon or rectum with stage IV (metastatic) liver-only disease, as defined by staging with CT scans.
2. Patients must have a baseline evaluation to determine whether liver metastases are resectable (e.g. a single liver metastasis in a resectable location)or unresectable (surgical consultation is recommended). Both groups are eligible for this study.
3. Tumor tissue must reveal wild-type KRAS expression (i.e. no KRAS mutation) prior to study entry (see Section 7.4.4.).
4. Patients must have at least one unidimensional measurable lesion definable by CT scan. Disease must be measurable per RECIST version 1.1 criteria (see Section 9).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (see Appendix A).
6. Laboratory values as follows:

   ANC greater than 1500/μL

   Hgb greater than9 g/dL

   Platelets greater than 100,000/μL

   AST/SGOT less than 5.0 x ULN

   ALT/SGPT less than or equal to 5.0 x ULN

   Alk Phos less than or equal to 5.0 x ULN

   Bilirubin less than or equal to 1.5 x ULN

   Creatinine 1.5 mg/dL or calculated creatinine clearance 50 ml/min

   Magnesium LLN
7. Patient must have a life expectancy of greater than 12 weeks.
8. Patient must be greater than or equal to 18 years of age.
9. Patient must be accessible for treatment and follow-up.
10. Women of childbearing potential must have a negative serum or urine pregnancy test performed less than or equal to 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment and during the 6 months following completion of study treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
11. Patient must be able to understand the nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Prior systemic therapy for metastatic colorectal cancer (including chemotherapy, bevacizumab, cetuximab, panitumumab, and other targeted agents).
2. Adjuvant chemotherapy (and/or chemoradiation) for colorectal carcinoma ending less than or equal to 12 months prior to the diagnosis of metastatic cancer. Prior radiation therapy (in the metastatic setting) may be allowed if it was completed greater than or equal to 4 weeks prior to enrollment and measurable lesions are outside the radiation portal site.
3. Any detectable metastases in areas other than the liver.
4. Known liver disease or other significant medical illness that would exclude the patient as a candidate for resection of liver metastases.
5. Patients requiring therapeutic coumadin or heparin (for a history of pulmonary emboli or deep vein thrombosis [DVT]) will be excluded.
6. Patients who have had a major surgical procedure (not including mediastinoscopy), open biopsy, or significant traumatic injury less than or equal to 4 weeks prior to beginning treatment.
7. History of Gilbert's disease.
8. History of hypersensitivity to active or inactive excipients of any component of treatment (5 fluorouracil, irinotecan, panitumumab, and/or oxaliplatin), or known dipyrimidine dehydrogenase (DPD) deficiency
9. Serious cardiac arrhythmia requiring medication.
10. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, an infection requiring IV antibiotics, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Patient with known diagnosis of human immunodeficiency virus (HIV), hepatitis C virus or acute or chronic hepatitis B infection.
12. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
13. Use of any non-approved or investigational agent less than or equal to 28 days prior to administration of the first dose of study drug.
14. Past or current history of neoplasm other than the entry diagnosis with the exception of treated non melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a DFS greater than or equal to 5 years.
15. Patients with National Cancer Institute Common Terminology Criteria for Adverse Events v4.0 (NCI CTCAE) Grade 2 peripheral neuropathy.
16. Female patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, MD, Study Chair — SCRI Development Innovations, LLC
Locations (15):
- United States (15):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Hope Cancer Center, Terre Haute, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas

REFERENCES:
- [Derived] Bendell JC, Zakari A, Peyton JD, Boccia R, Moskowitz M, Gian V, Lipman A, Waterhouse D, LoCicero R, Earwood C, Lane CM, Meluch A. A Phase II Study of FOLFOXIRI Plus Panitumumab Followed by Evaluation for Resection in Patients With Metastatic KRAS Wild-Type Colorectal Cancer With Liver Metastases Only. Oncologist. 2016 Mar;21(3):279-80. doi: 10.1634/theoncologist.2015-0439. Epub 2016 Feb 24. PMID 26911408

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFOXIRI+Panitumumab Regimen: All patients will receive the FOLFOXIRI/panitumumab regimen, with drugs administered in the following order:
  * Panitumumab
  * Oxaliplatin
  * Irinotecan
  * Leucovorin
  * 5-Fluorouracil
  Panitumumab: 6 mg/kg, 60-90 minute IV infusion every 2 weeks
  Oxaliplatin: 85 mg/m2, 2-hour IV infusion every 2 weeks
  Irinotecan: 125 mg/m2, 1-hour IV infusion every 2 weeks
  Leucovorin: 200 mg/m2, 2-hour IV infusion every 2 weeks
  5-Fluorouracil: 3200 mg/m2 IV, 48-hour continuous infusion every two weeks
Period: Overall Study
Arm/Group | FOLFOXIRI+Panitumumab Regimen
Started | 15
Completed | 2 (Completed = patient is surgical candidate, underwent resection, received treatment to week 24.)
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: All patients on study
Arm/Group | FOLFOXIRI+Panitumumab Regimen
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 55 [39 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The Percentage of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Population: Includes all patients deemed to be evaluable for response who were evaluated for response
Measure: Number; unit: percentage of evaluable participants
Arm/Group | FOLFOXIRI+Panitumumab Regimen
Number analyzed (Participants) | 12
percentage of evaluable participants | 75

2. Secondary Outcome: R0 Resection Rate
Description: To determine the rate of complete (R0) resection for patients treated with this regimen.
Time Frame: 18 months
Population: Includes patients who were surgical candidates and underwent surgery on study
Measure: Number; unit: percentage of patients with surgery
Arm/Group | FOLFOXIRI+Panitumumab Regimen
Number analyzed (Participants) | 10
percentage of patients with surgery | 100

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 18 months
Population: All patients on study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOXIRI+Panitumumab Regimen
Number analyzed (Participants) | 15
months | 13.3 [4.2 to NA] — Upper bound of 95% confidence interval not reached at this time

4. Secondary Outcome: To Determine the Acute Toxicity Produced by This Regimen.
Description: The analyses of safety will be based on the frequency of adverse events and their severity for patients who received at least one dose of study treatment.
Time Frame: 18 months
Population: All patients on study
Measure: Number; unit: participants
Arm/Group | FOLFOXIRI+Panitumumab Regimen
Number analyzed (Participants) | 15
participants
  Rash | 12
  Diarrhea | 9
  Fatigue | 8
  Nausea | 8
  Mucositis | 7
  Peripheral neuropathy | 6
  Vomiting | 5
  Anorexia | 4
  Cold sensitivity | 4
  Constipation | 4
  Dehydration | 4
  Leukopenia | 4
  Anemia | 3
  Hypokalemia | 3
  Hypomagnesemia | 3
  Nail changes | 3
  Neutropenia | 3
  Taste alteration | 3
  Thrombocytopenia | 3
  Weight loss | 3
  Abdominal pain | 2
  Alopecia | 2
  Depression | 2
  Dizziness | 2
  Insomnia | 2
  Alkaline phosphatase increased | 1
  ALT increased | 1
  Anxiety | 1
  AST increased | 1
  Asthenia | 1
  Back pain | 1
  Blood bicarbonate increased | 1
  Decreased ejection fraction | 1
  Dry mouth | 1
  Dysesthesia | 1
  Dyspepsia | 1
  Edema | 1
  Epistaxis | 1
  Flashers | 1
  Hand-foot syndrome | 1
  Hematochezia | 1
  Hemorrhoids | 1
  Hyperpigmentation | 1
  Hypertension | 1
  Hypoalbuminemia | 1
  Hyponatremia | 1
  Infection - other | 1
  Infusion related reaction | 1
  Memory loss | 1
  Oral infection | 1
  Paraphasia | 1
  Pruritus | 1
  Speech impairment | 1
  Swollen tongue | 1

5. Secondary Outcome: Overall Survival (OS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 18 months
Population: All patients on study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOXIRI+Panitumumab Regimen
Number analyzed (Participants) | 15
months | NA [NA to NA] — Median overall survival and 95% confidence interval not reached at this time point - biostaticians are not reporting the lower bound of the 95% confidence interval when median overall survivial cannot be calculated

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | FOLFOXIRI+Panitumumab Regimen
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOXIRI+Panitumumab Regimen (N=15)
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOXIRI+Panitumumab Regimen (N=15)
Rash (Skin and subcutaneous tissue disorders) | 13
Diarrhea (Gastrointestinal disorders) | 11
Fatigue (General disorders) | 9
Mucositis (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 6
Peripheral Sensory Neuropathy (Nervous system disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
White Blood Cell Decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 5
General disorders and administration site conditions - Other, cold sensitivity (General disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Neutrophil Count Decreased (Investigations) | 4
Platelet Count Decreased (Investigations) | 4
Abdominal Pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 3
Anemia (Blood and lymphatic system disorders) | 3
Anxiety (Psychiatric disorders) | 3
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 3
Weight loss (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 2
Chills (General disorders) | 2
Depression (Psychiatric disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dysesthesia (Nervous system disorders) | 2
Fever (General disorders) | 2
Gastrointestinal disorders - Other, bloody stools (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 2
Nervous system disorders - Other, speech impairment (Nervous system disorders) | 2
Rectal Pain (Gastrointestinal disorders) | 2
Upper Respiratory Infection (Infections and infestations) | 2
Alkaline phosphatase increased (Investigations) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Blurred vision (Eye disorders) | 1
Burn (Injury, poisoning and procedural complications) | 1
Conjunctivitis (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dry eye (Eye disorders) | 1
Edema limbs (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Eye disorders - Other, blepharitis (Eye disorders) | 1
Flashing lights (Eye disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, enlarged tongue (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, stomatitis (Gastrointestinal disorders) | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Gum infection (Infections and infestations) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infections and infestations - Other, pneumonia (Infections and infestations) | 1
Infections and infestations - Other, unknown (Infections and infestations) | 1
infusion related reaction (General disorders) | 1
Investigations - Other, blood bicarbonate decreased (Investigations) | 1
Investigations - Other, blood bicarbonate increased (Investigations) | 1
Joint infection (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Memory impairment (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Paronychia (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, acute renal insufficiency (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites